CLINICAL TRIAL: NCT01495507
Title: Cross-cultural Adaptation and Validation of the German Version of the Kujala Score in Patients With Patellofemoral Instability - a Prospective Multi-centric Study
Brief Title: Validation of Kujala German
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Michael Liebensteiner, MD, PhD, Medical University Innsbruck
Other Study IDs: Kuj-Germ-1
Record Dates: First submitted 2011-12-19; First posted 2011-12-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Validation of Kujala Score German Version in Patients With Patellofemoral Instability and Scheduled MPFL-reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patellofemoral Instability: Patients with diagnosis of patellofemoral instability receiving MPFL-reconstruction as part of the clinical routine
  Interventions: Procedure: MPFL- Reconstruction

INTERVENTIONS:
Procedure: MPFL- Reconstruction

SUMMARY:
The field of patellofemoral disorders and accordant therapeutical interventions is a high turnover research field. It is important to verify the clinical outcome with appropriate measuring tools. There is evidence that the Kujala score is a reliable and widely used measuring instrument of patellofemoral disorders. Indeed, the Kujala score was already used in many studies investigating patellofemoral disorders - also in german speaking patient groups. Unfortunately, we are not aware of a validated german version of the Kujala score. Other relevant knee outcome scores were already successfully translated into german language and validated by previous investigators.

So, it is the aim of our study to cross-culturally adapt and then to validate the Kujala score for use in German-speaking individuals with patellofemoral instability. It is hypothesized that the german version of the Kujala score shows:

* High divergent construct validity as determined by significant differences between patients and controls (hypothesis 1)
* High convergent construct validity as determined by significant correlations with other relevant scoring systems (hypothesis 2)
* High reliability (hypothesis 3)
* High responsiveness (hypothesis 4)

ELIGIBILITY:
Inclusion Criteria:

* german speaking
* MPFL-reconstruction planed

Exclusion Criteria:

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with patellofemoral instability & scheduled MPFL-reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Kujala Score | 1 year
KOOS (Knee Injury and Osteoarthritis Outcome Score) | 1 year
Marx Activity Scale | 1 year
SF-12 (Short - Form 12) | 1 year
VAS pain | 1 year
Lysholm Score | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. Orthop. Surgery, Medical Univ. Innsbruck, Innsbruck, Tyrol, Austria